CLINICAL TRIAL: NCT04427046
Title: Clinical Presentation and Outcome of Acute Myocardial Infarction in Native Versus Non-native Young Population in Saudi Arabia
Brief Title: Acute Myocardial Infarction in Native Versus Non-native Young Population in Saudi Arabia
Acronym: YAMI
Status: Completed | Type: Observational
Sponsor: Saud Al Babtain Cardiac Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SBCC-2018-14
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Acute Myocardial Infarction
Keywords: Young; Saudi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A retrospective study collecting the data of young patients admitted with diagnosis of Acute Myocardial Infarction.

DETAILED DESCRIPTION:
A retrospective study investigating young adults aged <45 years for males and <55 years for females admitted at Saud Al Babtain Cardiac Center with diagnosis of Acute Myocardial Infarction, determining its risk factors for Coronary Artery Disease (CAD) related to cultural characteristics and common positive consanguinity of parents as well as the prevalent diabetes and smoking.

ELIGIBILITY:
Inclusion Criteria:

* <45 years old for male and <55 years old for female
* patients admitted with diagnosis of Acute Myocardial Infarction

Exclusion Criteria:

* <17 and >55 years old male and female
* patients admitted with diagnosis other than Acute Myocardial Infarction.

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young adults, saudi or non-saudi, with Acute Myocardial Infarction.
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Number of young adults hospitalized with primary diagnosis of Acute Myocadial Infarction. | 2 years
  Clinical Presentation and Outcome of Acute Myocardial Infarction in Native Versus Non-native Young Population in Saudi Arabia

CONTACTS AND LOCATIONS:
Overall Officials: Ali Youssef, MD, Principal Investigator — Saud Al Babtain Cardiac Center
Locations (1):
- Saud Al Babtain Cardiac Center, Dammam, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided